CLINICAL TRIAL: NCT06679881
Title: A Long-term, Open-label Study to Evaluate the Safety and Efficacy of Orally Administered Deucrictibant Extended-Release Tablet for Prophylaxis Against Angioedema Attacks in Adolescents and Adults With Hereditary Angioedema
Brief Title: Long-Term, Open-label Study of Oral Deucrictibant Extended-Release Tablet for Prophylaxis Against Angioedema Attacks in Adolescents and Adults With HAE
Acronym: CHAPTER-4
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pharvaris Netherlands B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHA022121-C307
Record Dates: First submitted 2024-10-24; First posted 2024-11-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Hereditary Angioedema (HAE)
Keywords: HAE; Oral Treatment; Bradykinin B2 Receptor Antagonists; PHVS719; PHA121; Deucrictibant; Prophylaxis
MeSH Terms: conditions — Angioedemas, Hereditary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Deucrictibant (Experimental): Deucrictibant
  Interventions: Drug: Deucrictibant

INTERVENTIONS:
Drug: Deucrictibant — Deucrictibant extended-release tablet for once daily oral use

SUMMARY:
This is a Phase 3, multicenter, long-term, open-label study to evaluate the safety and efficacy of once-daily orally administered deucrictibant extended-release tablet for prophylaxis to prevent angioedema attacks in participants aged ≥12 years with Hereditary Angioedema

DETAILED DESCRIPTION:
The study consists of a Screening Period during which eligibility is confirmed (only for participants not rolling over within 28 days from a previous deucrictibant prophylactic study), a Treatment Period in which participants will receive open-label deucrictibant extended-release tablet once daily for approximately 130 weeks, followed by an End of Study visit after maximum 4 weeks. Participants will undergo regular safety (e.g. lab draws) and efficacy assessments, will complete an electronic diary daily, and also complete questionnaires at predefined timepoints during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent/assent.
2. Male or female, aged ≥12 years at the time of providing written informed consent/assent.
3. Diagnosis of hereditary angioedema (HAE)
4. For participants that did not participate in a previous deucrictibant prophylactic study: history of at least 1 attack in the last 3 consecutive months prior to Screening
5. Reliable access and ability to use standard of care on-demand treatments to effectively manage acute HAE attacks.
6. Willing and able to adhere to all protocol requirements, including eDiary and ePRO data recording.
7. Female participants of childbearing must agree to the protocol specified pregnancy testing and contraception methods.

Exclusion Criteria:

1. Any diagnosis of angioedema other than HAE
2. Participation in a clinical study with any other investigational drug within the last 30 days or within 5 half-lives of the investigational drug at ICF signature (whichever is longer)
3. Prior gene therapy for any indication at any time
4. Participants who discontinued from previous studies with deucrictibant prophylactic and/or on-demand treatment due to safety reasons or compliance issues that, in the opinion of the Investigator, would interfere with the participant's safety or compliance to participate in the study
5. Exposure to ACE inhibitors or any estrogen-containing medications with systemic absorption within 4 weeks of Screening
6. Use of prophylactic treatment for HAE within 2 weeks of Screening for C1INH, oral kallikrein inhibitors, or anti-fibrinolytics; within 4 weeks of Screening for attenuated androgens; within 5 half-lives of Screening for monoclonal antibodies, or within 7 days of Screening for short-term prophylaxis
7. Any females who are pregnant, plan to become pregnant, or are currently breast-feeding
8. Abnormal hepatic function
9. Moderate or severe renal impairment
10. Any clinically significant comorbidity or systemic dysfunction that would interfere with the participant's safety or ability to participate in the study.
11. History of alcohol or drug abuse within the previous year, or current evidence of substance dependence or abuse
12. Use of medications that are moderate and strong inhibitors or strong inducers of CYP3A4 within the last 30 days or within 5 half-lives (whichever is longer) of the time of randomization
13. Known hypersensitivity to deucrictibant or any of the excipients of the study drug

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse events (TEAEs), including serious adverse events (SAEs), adverse events of special interest (AESIs), and TEAEs leading to study drug discontinuation | Up to 138 weeks
Change in heart rate | Up to 138 weeks
Change in blood pressure | Up to 138 weeks
Change in body temperature | Up to 138 weeks
Change in clinical laboratory tests from baseline | Up to 138 weeks
  Hematology, blood chemistry, and urinalysis. Descriptive in nature, no formal statistical hypothesis testing will be performed.
Change in electrocardiograms (ECGs) from baseline | Up to 138 weeks
  Digital triplicate 12-lead ECG. Descriptive in nature, no formal statistical hypothesis testing will be performed.

SECONDARY OUTCOMES:
Time-normalized number of Investigator-confirmed HAE attacks during the Treatment Period | 130 weeks
Time-normalized number of Investigator-confirmed HAE attacks treated with on-demand medication during the Treatment Period | 130 weeks
Time-normalized number of Investigator-confirmed moderate or severe HAE attacks during Treatment Period | 130 weeks
Time-normalized number of Investigator-confirmed severe HAE attacks during the Treatment Period | 130 weeks
Proportion of time without angioedema symptoms during the Treatment Period | 130 weeks
Patient reported outcome: Angioedema Quality of Life (AE-QoL) questionnaire | 130 weeks
  The AE-QoL is a short 17-item questionnaire designed to retrospectively assess HRQoL, with a recall period of 4 weeks. Its results can be displayed as a total score or as 4 domain scores. The scores range from 0 to 100, after linear transformation of raw values, with higher scores indicating higher HRQoL impairment.
Patient reported outcome: Patient Global Assessment of Change (PGA-Change) | 130 weeks
  PGA-Change assesses on a 5-point scale how the participant's QoL has been impacted by HAE since start taking the study drug.
Patient reported outcome: Angioedema Control Test 4-week version (AECT-4wk) | 130 weeks
  AECT-4wk measures disease control retrospectively, it comprises 4 questions over a 4-week recall period. Scores for the responses in the AECT range from 0 to 16, with higher scores indicating better disease control (≤ 9 poorly controlled; ≥ 10 well controlled).
Patient reported outcome: Work Productivity and Activity Impairment Questionnaire - Specific Health Problem (WPAI-SHP) | Up to 134 weeks
  WPAI-SHP is a questionnaire assessing how a health condition impacts a person's ability to work and do regular activities and it includes 4 domains. Scores indicate the percentage of time the patient missed work or was less productive owing to HAE-related complications.
Patient reported outcome: Abbreviated Treatment Satisfaction Questionnaire for Medication (TSQM-9) | Up to 134 weeks
  TSQM-9 is a 9-item questionnaire evaluating patient treatment satisfaction and it includes 3 domains. Scoring is by domain and each domain score is computed by summing the individual TSQM items in each domain and then transforming the composite score into a value ranging from 0 to 100, with higher scores indicating higher satisfaction.
Pharmacokinetics [PK]: Deucrictibant plasma concentration pre-dose (Ctrough) | 130 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Pharvaris, Study Director — Pharvaris Netherlands B.V.
Locations (23):
- United States (3):
  - Study Site, Santa Monica, California
  - Study Site, Walnut Creek, California
  - Study Site, St Louis, Missouri
- Australia (2):
  - Study Site, Melbourne
  - Study Site, Perth
- Study Site, Vienna, Austria
- Study Site, Sofia, Bulgaria
- Study Site, Montreal, Canada
- Germany (2):
  - Study Site, Berlin
  - Study Site, Frankfurt
- Study Site, Hong Kong, Hong Kong
- Study Site, Dublin, Ireland
- Study Site, Padua, Italy
- Study Site, Krakow, Poland
- Study Site, Cape Town, South Africa
- South Korea (2):
  - Study Site, Daegu
  - Study Site, Seoul
- Study Site, Barcelona, Spain
- United Kingdom (5):
  - Study Site, Brighton
  - Study Site, Bristol
  - Study Site, Cambridge
  - Study Site, London
  - Study Site, Plymouth